CLINICAL TRIAL: NCT03404687
Title: Comparative Study Between Use of the Risk of Malignancy Index Versus Assiut Scoring Model in Preoperative Prediction of Adnexal Malignancy
Brief Title: Risk of Malignancy Index and Assiut Scoring Model for Adnexal Malignancy
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Other Study IDs: RMI_ASS
Record Dates: First submitted 2018-01-13; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Risk Malignant Index
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with adnexal masses
  Interventions: Radiation: ultrasound; Diagnostic Test: cancer antigen 125 level; Radiation: Doppler

INTERVENTIONS:
Radiation: ultrasound — for assessment of adnexal masses size and pattern
Diagnostic Test: cancer antigen 125 level — for prediction of malignancy
Radiation: Doppler — for detection of blood flow

SUMMARY:
The presence of an adnexal mass is a frequent reason for a woman to be referred to a gynaecologist. The discrimination between benign and malignant adnexal masses is central to decisions regarding clinical management and surgical planning in such patients. Patients with malignant tumours should be referred to a gynaecological oncologist, as the quality of cytoreductive surgery and surgical staging/lymph node dissection are important prognostic factors in ovarian cancer. These specialized surgical procedures require the specific skills and experience provided by gynaecologic oncology surgeons. Furthermore, appropriate and timely referral to a gynaecologic oncologist has been proven to increase survival in patients with ovarian cancer.Conversely, patients believed to have a benign mass requiring surgery are able to have this performed by a general gynaecologist. A standardized method for preoperative identification of probable malignant masses would allow optimization of first-line treatment for women with ovarian cancer. A risk of malignancy index would be valuable for the selective referral of relevant patients to specialized oncology centres. Currently, clinical examination, ultrasound assessment, and assays of tumour markers are part of the standard work-up for an adnexal mass. Although none of these indicators alone is very sensitive or specific for detecting malignancy, an index developed by Jacobs et al. incorporates information about the patient's menopausal status and serum Cancer antigen A-125 levels, and ultrasound characteristics of the mass to predict the risk of malignancy with greater sensitivity and specificity than any one factor alone.Some of the potential advantages of risk malignant index include rapid triage of patients through the referral system and fewer operations for benign masses being performed by gynaecologic oncologists.

ELIGIBILITY:
Inclusion Criteria:

1. Age at menarche to 60 years.
2. Presence of ovarian mass clinically by vaginal or bimanual examination.
3. Presence of sonographically diagnosed ovarian mass.
4. Accepting and signing the informed written consent.

Exclusion criteria

1. Known diagnosis of nature of mass by previous biopsy or ovarian malignancy scheduled for second look operation.
2. Patient unfit for surgery or inoperable.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients has any adnexal mass by ultrasound
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Number of women has a malignant adnexal mass | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided